CLINICAL TRIAL: NCT02047942
Title: A Randomized Controlled Trial Comparing Home-based Training With Telemonitoring Guidance Versus Center-based Cardiac Rehabilitation in Patients With Coronary Heart Disease: the TRiCH-study
Brief Title: Telerehabilitation in Coronary Heart Disease
Acronym: TRiCH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: KU Leuven (Other)
Collaborators: Jessa Hospital (Other); Hasselt University (Other)
Responsible Party: Principal Investigator, Véronique Cornelissen, Dr, KU Leuven
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MOVE-AGE_09_2013
Record Dates: First submitted 2014-01-27; First posted 2014-01-28 (Estimated); Last update posted 2019-06-24 (Actual); Status verified 2019-06

CONDITIONS: Coronary Artery Disease (CAD) (E.G., Angina, Myocardial Infarction, and Atherosclerotic Heart Disease (ASHD)); Myocardial Infarction; Percutaneous Transluminal Cutting Balloon Angioplasty of Popliteal Vein Using Fluoroscopic Guidance
MeSH Terms: conditions — Coronary Artery Disease; Angina Pectoris; Myocardial Infarction

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Center-based cardiac rehabilitation (Active Comparator): Patients randomized to the center-based training group will continue their training sessions at the outpatient clinics of UZ Leuven under direct supervision of physical therapists
  Interventions: Behavioral: Center-based cardiac rehabilitation
- Home-based training with telemonitoring guidance (Experimental): Patients will receive an patient-tailored exercise prescription and will be asked to perform the exercise sessions in their home environment wearing heart rate monitors. Training data will be accessed by the research group on weekly basis in order to keep a record of frequency; duration and intensity of the sessions. Feedback will be given weekly to every patient.
  Interventions: Behavioral: Home-based training with telemonitoring guidance
- Control (No Intervention)

INTERVENTIONS:
Behavioral: Center-based cardiac rehabilitation
  Arms: Center-based cardiac rehabilitation
Behavioral: Home-based training with telemonitoring guidance
  Arms: Home-based training with telemonitoring guidance

SUMMARY:
Cardiovascular diseases are the main cause of death worldwide. Aerobic fitness is related to long-term survival and a reduction in mortality and recurrent nonfatal myocardial infarction in subjects with cardiovascular disease. However, the majority of cardiac patients do not engage in enough physical activity to obtain benefits or in the long-term struggle to maintain a physically active lifestyle. There is a need for innovative rehabilitation methods aiming at increasing longer-term adherence and hence more sustained effects on health related physical fitness. One strategy might be the use of home-based training in combination of telemonitoring guidance. Therefore, the main objective of this randomized controlled clinical trial is to compare the longer-term (=1 year) effects of a 3-month supervised center-based rehabilitation program with a patient-tailored home-based cardiac rehabilitation program with telemonitoring guidance in CAD patients (phase III). The primary outcome measure is physical fitness. It is hypothesized that patients randomized to a home-based training program with telemonitoring guidance will demonstrate higher levels of physical activity at one year of follow-up, resulting in higher levels of physical fitness, compared to patients who have been enrolled to the supervised center-based cardiac rehabilitation program or control group. Ninety patients will be randomized to Home-based training, a center-based cardiac rehabilitation program or an advice only group (= control group). Assessment will be performed at baseline, immediately at completion of the intervention and at one-year of follow-up and will include measurements of exercise tolerance, cardiovascular risk factors, physical activity, muscle strength, endothelial function, health-related quality.

ELIGIBILITY:
Inclusion Criteria:

* Patients with CAD (post-PCI, post-MI, post-CABG)
* Patients on optimal medical treatment and stable with regard to symptoms and pharmacotherapy for at least 6 weeks
* Patients have successfully completed the 3 month ambulatory cardiac rehabilitation in hospital program
* 39 yrs < age < 76 years
* access to internet facilities or PC at home

Exclusion Criteria:

* Significant undercurrent illness last 6 weeks
* Known severe ventricular arrhythmia with functional or prognostic significance; significant myocardial ischemia, hemodynamic deterioration or exercise-induced arrhythmia at screening or heart disease that limits exercise
* Co-morbidity that may significantly influence one-year prognosis
* Functional of mental disability that may limit exercise

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2014-02 (Actual); Primary Completion 2017-08 (Actual); Study Completion 2017-08 (Actual)

PRIMARY OUTCOMES:
exercise tolerance | 1 year
  comparison of evolution of exercise tolerance from baseline to one-year
exercise tolerance | 12 weeks
  comparison of evolution of exercise tolerance from baseline to 12 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- KU Leuven, Leuven, Belgium

REFERENCES:
- [Derived] Avila A, Claes J, Buys R, Azzawi M, Vanhees L, Cornelissen V. Home-based exercise with telemonitoring guidance in patients with coronary artery disease: Does it improve long-term physical fitness? Eur J Prev Cardiol. 2020 Mar;27(4):367-377. doi: 10.1177/2047487319892201. Epub 2019 Dec 1. PMID 31787026
- [Derived] Avila A, Claes J, Goetschalckx K, Buys R, Azzawi M, Vanhees L, Cornelissen V. Home-Based Rehabilitation With Telemonitoring Guidance for Patients With Coronary Artery Disease (Short-Term Results of the TRiCH Study): Randomized Controlled Trial. J Med Internet Res. 2018 Jun 22;20(6):e225. doi: 10.2196/jmir.9943. PMID 29934286